CLINICAL TRIAL: NCT02533739
Title: Impact Des déficits Vestibulaires Sur le développement Des Fonctions Visuo-spatiales.
Brief Title: Vestibular Disorder and Visuo-spatial Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/28MAR/143
Record Dates: First submitted 2015-08-12; First posted 2015-08-27 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Vestibular Diseases; Vertigo
MeSH Terms: conditions — Vestibular Diseases; Vertigo

ARMS (2):
- Patient group (Experimental): This group will consist of vestibular patients and/or participants with vertigo.
  Interventions: Behavioral: Cognitive and neuropsychological assesment
- Control group (Sham Comparator): This group will consist of participants without vestibular/vertigo impairments.
  Interventions: Behavioral: Cognitive and neuropsychological assesment

INTERVENTIONS:
Behavioral: Cognitive and neuropsychological assesment

SUMMARY:
The purpose of these studies is to determine whether vestibular disorders could affect visuo-spatial cognition. Visuo-spatial cognition will be evaluated using a new questionnaire and a new computerized test using a digital tablet in different studies.

ELIGIBILITY:
For participants of the questionnaire study :

Participants with vertigo complaints versus participants without vertigo complaints.

For patients of the behavioural study :

Inclusion Criteria:

* Vestibular disorder (with or without vertigo)
* Deafness / hard of hearing

Exclusion Criteria:

* Neurological or psychiatric conditions
* Cochlear Implant (for functional magnetic resonance imaging study)

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Vestibular questionnaire (Newly developed to evaluate cognitive abilities) | Within one week after recruitment
  Participants will be recruited and tested within one week of recruitment. Testing will be online and will take around 20 minutes on average. The new questionnaire will evaluate demographic questions, and different cognition abilities using a likert-scale.
Standard computerized cognitive assessment (For example : Test of attentional performance, digit span, visuo-spatial span, line bisection task,...) | Within one week after recruitment
  Participants will be recruited and tested within one week of recruitment. Testing will be at the hospital and will take 2 hours maximum. Standard computerized cognitive assessment will be used such as the Test of attentional performance (TAP2.2), digit span, visuo-spatial span, line bisection task, etc. Reaction times, errors and omissions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Naïma Deggouj, Study Director — Cliniques universitaires Saint-Luc-UCL
Locations (1):
- Cliniques universitaires Saint-Luc-UCL, Brussels, Belgium